CLINICAL TRIAL: NCT02077361
Title: An Open Label Clinical Trial of Retinal Gene Therapy for Choroideremia Using an Adeno-associated Viral Vector (AAV2) Encoding Rab-escort Protein-1 (REP1)
Brief Title: An Open Label Clinical Trial of Retinal Gene Therapy for Choroideremia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Canada Foundation for Innovation (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Choroideremia Research Foundation Canada (Unknown); Foundation Fighting Blindness (Other); Imperial College London (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00028599; File # 9427-U0180-84C (Other: Health Canada)
Record Dates: First submitted 2014-02-26; First posted 2014-03-04 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Choroideremia
Keywords: choroideremia; gene therapy; gene transfer
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental): Patients will receive a subretinal injection of 0.10 ml of the rAAV2.REP1 vector drug substance. It is a colourless opalescent frozen liquid with no visible particles. Each patient will be given a one-time dose in one eye.
  It is the same vector used in the United Kingdom Phase I/II trial logged at: http://clinicaltrials.gov/ct2/show/NCT01461213.
  Interventions: Genetic: rAAV2.REP1 vector

INTERVENTIONS:
Genetic: rAAV2.REP1 vector — No additional details needed.

SUMMARY:
A project has been developed in Edmonton, Alberta, Canada to enable male patients with choroideremia to access a clinical trial that replaces the defective gene with a normal copy. This experiment is designed to show that the transfer of a normal copy of the gene to the eye is not only safe but may improve the sight of patients. Only Canadian subjects who meet criteria will be recruited.

DETAILED DESCRIPTION:
This is an open label study involving a total of 6 male patients. Screening and patient medical records will determine patient eligibility. Patients will receive a subretinal injection of the rAAV2.REP1 vector by a trained vitreoretinal surgeon in one eye. Each patient will be followed up for 24 months after treatment to assess the primary and secondary endpoints of this study using a number of outcome measures. However, further follow-up will continue after the study on an annual basis for a minimum of ten years. Data will continue to be analyzed by members of the study group after this study is complete.

ELIGIBILITY:
Inclusion Criteria:

* The research subject is willing and able to give informed consent for participation in the study.
* Male aged 18 years or above.
* Diagnosed with choroideremia (with genotyping or evidence of lack of the gene product with immunohistochemistry) and in good health.
* Active degeneration of the retina (the expectation of significant decline in visual function without any intervention over the subsequent 5 years) with OCT (optical coherent tomography) changes visible within the macula.
* Willingness to allow his general physician and ophthalmologist, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply.

* Female or child research subject (under the age of 18).
* Men unwilling to use barrier contraception methods, if relevant.
* Previous history of retinal surgery or ocular inflammatory disease (uveitis).
* Grossly asymmetrical retinal disease or other ocular morbidity which might confound adopting the fellow eye as a long-term comparator.
* Any other significant systemic disease or disorder which, in the opinion of the investigator, may either put the research subject at risk because of participation in the study, or may influence the result of the study, or the research subject's ability to participate in the study. This would include a contraindication to oral prednisolone, such as a history of gastric ulcer).
* Research subjects who have participated in another research study involving an investigational product within the past year.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08-30 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with ocular and systemic adverse events | 2 years
  This is assessed by standard ocular examinations and vector dissemination and inflammation assays.

SECONDARY OUTCOMES:
Changes in visual field | Baseline and up to 2 years following vector delivery
  This is assessed by Goldmann perimetry and microperimetry; measurements before and after vector delivery are compared.
Changes in visual function | Baseline and 2 years following vector delivery
  This is assessed by multifocal electrophysiology, full field scotopic threshold, spectral domain optical coherent tomography, fundus photography and fundus autofluorescence; measurements before and after vector delivery are compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M MacDonald, MD, CM, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Background] Hauswirth WW, Aleman TS, Kaushal S, Cideciyan AV, Schwartz SB, Wang L, Conlon TJ, Boye SL, Flotte TR, Byrne BJ, Jacobson SG. Treatment of leber congenital amaurosis due to RPE65 mutations by ocular subretinal injection of adeno-associated virus gene vector: short-term results of a phase I trial. Hum Gene Ther. 2008 Oct;19(10):979-90. doi: 10.1089/hum.2008.107. PMID 18774912
- [Background] Bainbridge JW, Smith AJ, Barker SS, Robbie S, Henderson R, Balaggan K, Viswanathan A, Holder GE, Stockman A, Tyler N, Petersen-Jones S, Bhattacharya SS, Thrasher AJ, Fitzke FW, Carter BJ, Rubin GS, Moore AT, Ali RR. Effect of gene therapy on visual function in Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2231-9. doi: 10.1056/NEJMoa0802268. Epub 2008 Apr 27. PMID 18441371
- [Background] Bennicelli J, Wright JF, Komaromy A, Jacobs JB, Hauck B, Zelenaia O, Mingozzi F, Hui D, Chung D, Rex TS, Wei Z, Qu G, Zhou S, Zeiss C, Arruda VR, Acland GM, Dell'Osso LF, High KA, Maguire AM, Bennett J. Reversal of blindness in animal models of leber congenital amaurosis using optimized AAV2-mediated gene transfer. Mol Ther. 2008 Mar;16(3):458-65. doi: 10.1038/sj.mt.6300389. Epub 2008 Jan 22. PMID 18209734
- [Background] MacLaren RE. An analysis of retinal gene therapy clinical trials. Curr Opin Mol Ther. 2009 Oct;11(5):540-6. PMID 19806502
- [Background] MacLaren RE, Groppe M, Barnard AR, Cottriall CL, Tolmachova T, Seymour L, Clark KR, During MJ, Cremers FP, Black GC, Lotery AJ, Downes SM, Webster AR, Seabra MC. Retinal gene therapy in patients with choroideremia: initial findings from a phase 1/2 clinical trial. Lancet. 2014 Mar 29;383(9923):1129-37. doi: 10.1016/S0140-6736(13)62117-0. Epub 2014 Jan 16. PMID 24439297
- [Derived] Brooks SP, Benjaminy S, Bubela T. Participant perspectives on a phase I/II ocular gene therapy trial (NCT02077361). Ophthalmic Genet. 2019 Jun;40(3):276-281. doi: 10.1080/13816810.2019.1630843. Epub 2019 Jul 4. PMID 31269854
- See also: Choroideremia Overview — http://ffb.ca/learn/eye-diseases/